CLINICAL TRIAL: NCT01065207
Title: ANRS HIV CONTROLLERS NATIONAL OBSERVATORY
Brief Title: Patients Infected With HIV Since More Than 10 Years With a Plasma Viral RNA <400 Copies / mL in the Absence of Any Treatment: Study Mechanisms Involved in Controlling the Infection
Acronym: ANRS CO18
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 05-0222
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient (No Intervention)
  Interventions: Biological: blood test at day one

INTERVENTIONS:
Biological: blood test at day one — Epidemiological, clinical, virological, and immunological data will be collected.
  Clinical events as neoplasia will be collected

SUMMARY:
The investigators have previously described a limited group of HIV-1-infected patients, we called HIV controllers (HIC), who have been infected for more than 10 years, in whom viral replication is spontaneously controlled without any treatment. These patients are defined according to virological criteria: more than 90% of the quantifications of plasma viral load should be less than 400 RNA copies/mL. The purpose of the ANRS EP36 study was to characterize these patients.

DETAILED DESCRIPTION:
To study the virological and immunological features of these patients, a consortium of research teams has been set up. Several results were obtained (cf publications) : HIC are infected with replication-competent virus, HIV infects HIC CD4 T cells ex vivo but the CD8 T cells fully control this viral replication. This study led to set up a national observatory of the HICs. This observatory, set up from May 2006 to May 2008, has allowed to identify and include 86 HIC patients in France (about one hundred had been reported by the ANRS centers). When a patient is included, clinical data are collected and a biologic collection set up which can be used in genomic studies. The main characteristics of the patients included in the observatory are a median age at the diagnosis of HIV infection of 29 years (range 1-49), a median age at inclusion of 45 years [19-78], 42% are women, 87% are caucasians. The median year of HIV diagnosis is 1989 (1983-1999), so a median of 18 years of known HIV infection. The CD4 median between 1986 and 2008 is 762 CD4/mm3 [IQR:589-962], 3% of the 1368 measures are ≤ 350 /mm3; 23% patients have a CD4 T cell count < 500/mm3 and 6% < 350/mm3 at the inclusion consultation. The CD4 slope on this period shows a slow decrease estimated to -13 [-15,-11] CD4/mm3 per year. Between 1989 and 2007, 2% of the viral loads measured were ≥ 1000 RNA copies/mL. The viral load at inclusion is > 400 RNA copies/mL in 4%. Median viral DNA at the inclusion in the observatory is 1, 75 [1, 44-2, 07] log copies/millions PBMC.

The transformation of the observatory in a cohort CO 18 has several goals. The first one is to allow the long-term follow-up of the HIV controllers. Epidemiological, clinical, virological, and immunological data will be collected. The outcome of these patients is a major question: some patients could loose their HIC status either because of a drop in their CD4 T cell counts to a level below 200/mm3 without major viral replication or because viral replication becomes detectable. To understand the mechanisms involved in the control of the viral replication in HIC implies to study the patients in whom the viral control is lost and to compare them to the HIC in whom the control is preserved. Therefore it is of major importance to follow the patients now included in the observatory during a prolonged time. To increase the frequency of loss of control, the patients in whom the virus is controlled for at least 5 years but for less than 10 years will be included to increase the diversity of the HICs. Clinical events as neoplasias will be collected. The genomic studies will be continued with the benefits of new inclusions and european collaborations will be developed. The question of the quality-of-life of the patients HIC will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* able to give written consent
* who have been infected for more than 5 years
* not treated by ARV
* HIV positive serology
* Covered by French Social Security

Exclusion Criteria:

* Non compliance with the criteria of inclusion
* Pregnancy (inclusion can be postponed)
* Covered by French Social Security

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
to allow the long-term follow-up of the HIV controllers. Epidemiological, clinical, virological, and immunological data will be collected.

SECONDARY OUTCOMES:
To understand the mechanisms involved in the control of the viral replication in HIC implies to study the patients in whom the viral control is lost and to compare them to the HIC in whom the control is preserved

CONTACTS AND LOCATIONS:
Overall Officials: JP Faller, MD, Principal Investigator — CH Belfort; Pascal Roblot, PHD, Principal Investigator — CHU Poitiers; Gilles Beaucaire, MD, Principal Investigator — CHU Pointe à Pitre; Christine Rouger, MD, Principal Investigator — Hôpital Robert Debré REIMS; Jean Luc Delassus, MD, Principal Investigator — CHI Ballanger Aulnay sous Bois; Alain Devidas, MD, Principal Investigator — Hopital Gilles De Corbeil Corbeil; Louis Bubertet, Principal Investigator — Hopital St Louis Paris; Michèle Bentata, MD, Principal Investigator — Hopital Avicenne BOBIGNY; Alexandra Compagnucci, MD, Principal Investigator — Hopital Hotel Dieu Paris; Philippe Genet, PHD, Principal Investigator — Hopital Victore Dupouy Argenteuil; Olivier Patey, PHD, Principal Investigator — CHI Villeneuve St Goerges; Marie Christine Drobacheff, MD, Principal Investigator — CHU St Jacques Besancon; Helder Gil, MD, Principal Investigator — CHU Minjoz Besanson; Eric Oksenhendler, PHD, Principal Investigator — Hopital St Louis Paris; Frédéric Lucht, PHD, Principal Investigator — Hopital Bellevue St Etienne; Michel Dupon, PHD, Principal Investigator — Hopital Pellegrin Bordeaux; Jean Luc Schmit, MD, Principal Investigator — Hôpital Nord Amiens; Daniel Sereni, PHD, Principal Investigator — St Louis ¨Paris; JP Viard, MD, Principal Investigator — Hotel Dieu Paris; JP Bru, MD, Principal Investigator — CH Annecy; JF Delfraissy, PHD, Principal Investigator — Le Kremlin Bicetre; Gilles Pichancourt, Principal Investigator — CH Henri Duffaut Avignon; André Pierre Blanc, MD, Principal Investigator — CH du payx d'Aix; Alain Lafeuillade, MD, Principal Investigator — Hopital Chalucet Toulon; Christophe Rapp, PHD, Principal Investigator — Hopital Inter Armées Bégin St Mandé; Pierre De Truchis, MD, Principal Investigator — Hopital Raymond Pointcarré Garches; Vincent Jeantils, MD, Principal Investigator — Hopital Jean Verdier Bondy; Daniel Vittecoq, PHD, Principal Investigator — Hopital Paul Brousse Villejuif; Gilles Pialoux, PHD, Principal Investigator — Hopital Tenon Paris; Olivier Bouchaud, PHD, Principal Investigator — Hopital Avicenne Bobigny; Francois Boué, PHD, Principal Investigator — Hopital Antoine Béclère Clamart; Laurence Weiss, PHD, Principal Investigator — HEGP Paris; Dominique Salmon Ceron, PHD, Principal Investigator — Cochin; Olivier Bletry, PHD, Principal Investigator — Hopital Foch Suresnes; Emmanuel Mortier, MD, Principal Investigator — Louis Mourier Paris; Alain Sobel, PHD, Principal Investigator — Hopital Henri Mondor Créteil; Christine Katlama, PHD, Principal Investigator — Pitié Salpétrière Paris; Anne Simon, MD, Principal Investigator — Pitié Salpétrière Paris; Pierre Marie Girard, PHD, Principal Investigator — St Antoine Paris; JM Molina, PHD, Principal Investigator — St Louis Paris; André Cabié, MD, Principal Investigator — Hopital Pierre Zobda Quitman Fort de France; JM Chennebault, MD, Principal Investigator — University Hospital, Angers; Philippe Morlat, PHD, Principal Investigator — Hopital St André Bordeaux; Pierre Weinbreck, PHD, Principal Investigator — CHU Limoges; JL Tourraine, PHD, Principal Investigator — Hopital Edouard Herriot - Lyon; Christian Trépo, PHD, Principal Investigator — Hopital Hotel Dieu Lyon; Isabelle Poizot Martin, MD, Principal Investigator — Ste Marguerite Marseille; Sophie Matheron, MD, Principal Investigator — Bichat Hospital; François Raffi, PHD, Principal Investigator — Hopital Hotel Dieu Nantes; Philippe Perré, MD, Principal Investigator — CH La Roche sur Yon; Pierre Delomonica, PHD, Principal Investigator — Hopital l'Archet Nice; Eric Rosenthal, PHD, Principal Investigator — Hopital l'Archet Nice; Christian Michelet, PHD, Principal Investigator — Rennes University Hospital; David Rey, MD, Principal Investigator — CHU Strasbourg; JM Besnier, PHD, Principal Investigator — Hopital Bretonneau Tours; Bruno Marchou, PHD, Principal Investigator — CHU Purpan (Toulouse); Renaud Verdon, PHD, Principal Investigator — Hopital de la côte de Nacre Caen; Christine Jacomet, MD, Principal Investigator — Hopital Hotel Dieu Clermont Ferrand; Lionel Piroth, MD, Principal Investigator — CHU Dijon; Pascale Leclercq, MD, Principal Investigator — Hopital Albet Michallon Grenoble; Yazdan Yazdanpanah, PHD, Study Director — Hopital Gustave Dron Tourcoing; Thierry May, PHD, Principal Investigator — Hopital de Brabois Nancy; Francois Caron, PHD, Principal Investigator — chu Rouen; Patrick Mercié, PHD, Principal Investigator — St André Bordeaux; Claire Series, PHD, Principal Investigator — Hopital Pellegrin Bordeaux; Philippe Granier, MD, Principal Investigator — CH Bourg en Bresse; Marc Gatfosse, MD, Principal Investigator — CH rené Arbeltier Coulomniers; Patrice Poubeau, MD, Principal Investigator — Groupe Hospitalier Sud Reunion St Pierre de la Réunion; Agnès Uludag, MD, Principal Investigator — Hopital Beaujon Clichy; Philippe Arsac, MD, Principal Investigator — CHR Orléans; Isabelle Delacroix, MD, Principal Investigator — CH intercommunal Créteil; Vincent Daneluzzi, MD, Principal Investigator — CASH Nanterre; Elisabeth Rouveix, MD, Principal Investigator — Hôpital Ambroise Paré Boulogne; Goerges Diab, MD, Principal Investigator — CH Noyon; Geneviève Berck Wirth, Principal Investigator — CH Mulhouse; Philippe Romand, MD, Principal Investigator — CHI Les hopitaux du Léman Thonon les Bains; Laurent Blum, MD, Principal Investigator — Hopital René Dubois Pontoise; Christophe Michau, MD, Principal Investigator — CH St Nazaire; Raymond Armero, MD, Principal Investigator — CHI Fréjus St Raphaël; Bernard Christian, MD, Principal Investigator — Hopital Notre Dame de Bon Secours Metz; Philippe Muller, MD, Principal Investigator — Hopital Beauregard Thionville; Henri Jardel, MD, Principal Investigator — CH Bretagne Atlantique Vannes; Elisabeth Carbonnel, MD, Principal Investigator — Hôpital Simone Weil Eaubonne; Laurent Hocqueloux, MD, Principal Investigator — Hopital La source Orléans; Marie Odile Lemaitre, MD, Principal Investigator — CH Juvisy sur Orge; Patrick Philibert, MD, Principal Investigator — Hopital Ambroise Paré Marseille; Paul Henry Consigny, MD, Principal Investigator — Institut Pasteur Paris; JM Ragnaud, PHD, Principal Investigator — Hopital Pellegrin Bordeaux; Daniel Garipuy, MD, Principal Investigator — Hopital Joseph Ducuing Toulouse; Beuscart MD Claude, Principal Investigator — CHU St Brieuc; Leprêtre MD Annie, Principal Investigator — Hôpital Simone Veil - Eaubonne; Duvivier MD Claudine, Principal Investigator — Institut Pasteur Paris; Garipuy MD Daniel, Principal Investigator — Hôpital Joseph Ducuing Toulouse; Aumaitre MD Hugues, Principal Investigator — Centre hospitalier de Perpignan; Rami MD Agathe, Principal Investigator — Lariboisière Paris; De Lavassière MD Marc, Principal Investigator — CH Général Montauban; Miailhes MD Patrick, Principal Investigator — Hôpital Croix Rousse Lyon
Locations (1):
- Le Kremlin-Bicêtre, France